CLINICAL TRIAL: NCT00310323
Title: Effect of Chronic Intermittent Nocturnal Hypoxia on Hepatic Drug Biotransformation in Children With Obstructive Sleep Apnea
Brief Title: Hepatic Drug Biotransformation in Children With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of Louisville (Other)
Responsible Party: Mary Jayne Kennedy, Pharm.D., Virginia Commonwealth University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSAS 003-03
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; phenotyping; cytochrome P450; drug metabolism; child
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Dextromethorphan; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Children with OSAS identified via sleep study
  Interventions: Drug: Dextromethorphan; Drug: Caffeine

INTERVENTIONS:
Drug: Dextromethorphan — 0.5 mg/kg (maximum 30 mg)
Drug: Caffeine — Administered as 4 ounces of Coca-Cola

SUMMARY:
The purpose of this research study is to determine the effect of chronic nighttime low oxygen saturations on selected body systems (liver) that break down drugs in children with obstructive sleep apnea syndrome (OSAS).

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of chronic intermittent nocturnal hypoxia on selected hepatic drug-metabolizing enzyme systems in children with OSAS. The specific aims are to evaluate the activities of cytochrome P450 (CYP)1A2, N-acetyltransferase-2 (NAT-2), xanthine oxidase (XO)and CYP2D6 in children with OSAS and to determine the effect of OSAS treatment on the activities of these enzyme systems.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 4 to 16 years with suspected uncomplicated OSAS

Exclusion Criteria:

* Children with complicated OSAS (craniofacial abnormalities, neuromuscular disorders)
* Children who are receiving medications known to induce or inhibit hepatic CYP1A2, NAT-2, XO, CYP2D6 or CYP3A4 activity
* Children who are exposed to second hand smoke for greater than 8 hours per day.
* Children with hypersensitivity to caffeine or dextromethorphan
* Children who are receiving corticosteroids or thyroid hormone

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2003-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Caffeine urinary molar ratio | Pre and post T&A
Dextromethorphan urinary molar ratio | Pre and post T&A

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jayne Kennedy, Pharm.D., Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - University of Louisville, Louisville, Kentucky
  - Virginia Commonwealth University, Richmond, Virginia